CLINICAL TRIAL: NCT06001203
Title: The Effect of Foot Reflexology on Pain, Walking Impairement and Ankle Brachial Index Level in Patients With Peripheral Artery Disease
Brief Title: Foot Reflexology and Pain and Ankle Brachial Index and Walking Impairement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Elif BUDAK ERTÜRK, Assistant Professor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KA23-152
Record Dates: First submitted 2023-08-03; First posted 2023-08-21 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): The intervention group is received two reflexology sessions.
  Interventions: Procedure: Reflexology
- control group (No Intervention): The control group is given routine care and no intervention will be performed.

INTERVENTIONS:
Procedure: Reflexology — Reflexology is a method that creates nervous, hormonal and energetic effects in the body using pressure, rubbing and stretching applied with special hand and finger techniques to reflex points corresponding to all parts, organs and systems of the body in the ears, hands and feet
  Arms: intervention group

SUMMARY:
This randomized controlled study aimed to determine the effect of foot reflexology on pain, walking impairement and ankle brachial index level in patients with peripheral artery disease

DETAILED DESCRIPTION:
Patients with PAH may experience pain in the legs, cramps, pain or aching symptoms (claudication) in the hip, thigh or leg calf, along with compulsive movements such as walking. Reflexology is reported to have effects such as protecting the tissue integrity of the feet, increasing skin turgor, reducing neuropathic pain and increasing peripheral blood flow. For this reason, this study aimed to determine the effect of foot reflexology on pain, walking impairement and ankle brachial index level in patients with peripheral artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years of age with PAH;
* no fractures or open wounds in both lower extremities;
* absence of unilateral or bilateral amputation of the lower extremities

Exclusion Criteria:

* having an acute infection with fever;
* requiring an acute surgical condition
* undergoing femoral-popliteal bypass surgery
* Having a verbal communication problem such as Alzheimer's or dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | Two reflexology sessions will be applied within one week and 4 measurements will be made. •Baseline (before first reflexology session), •After first reflexology session, •Before second reflexology session, •After second reflexology session
  Numeric Pain Rating Scale includes values ranging from 0 (no pain) - 10 (the worst pain)
Walking Impairment Questionnaire | Baseline, after 2 days second reflexology sessions
  The "Walking Impairment Questionnaire" is a self-report tool that evaluates walking distance and capacity. While the first 7 questions of the tool constitute the part where claudication and differential diagnosis are evaluated individually, the following 14 items are evaluated from 0 (can't do, very difficult) to 4 (no difficulty) on the Likert scale. The scale's walking distance, walking speed and stair climbing subscales are evaluated by evaluating the weights of each question, and total and subscale scores are calculated and evaluated between 0 and 100 points. A low score indicates poor walking performance.
Ankle Brachial Index | Two reflexology sessions will be applied within one week and 4 measurements will be made. •Baseline (before first reflexology session), •After first reflexology session, •Before second reflexology session, •After second reflexology session
  Ankle-brachial index is the ratio of the systolic blood pressure (SBP) measured at the ankle to that measured at the brachial artery.

SECONDARY OUTCOMES:
Toe oxygen saturation level | Two reflexology sessions will be applied within one week and 4 measurements will be made. •Baseline (before first reflexology session), •After first reflexology session, •Before second reflexology session, •After second reflexology session
  Toe oxygen saturation level is measured pulse oximetry. This method used to examine oxygen saturation in various parts of body.
Rate of Participants Edema level | Two reflexology sessions will be applied within one week and 4 measurements will be made. •Baseline (before first reflexology session), •After first reflexology session, •Before second reflexology session, •After second reflexology session
  Rate of Participants Edema level is measured from the ankle and calf with a tape measure.

CONTACTS AND LOCATIONS:
Overall Officials: Elif BUDAK ERTÜRK, PhD, RN, Principal Investigator — Baskent University Faculty of Health Science Department of Nursing
Locations (1):
- Baskent University, Ankara, Etimesgut, Turkey (Türkiye)